CLINICAL TRIAL: NCT01149499
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Valacyclovir 1000 mg Tablet and Valtrex Following a 1 x 1000 mg Dose in Healthy Subjects Under Fasting Conditions
Brief Title: Valacyclovir 1000 mg Tablet Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R04-1770
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Experimental): Test 1000 mg Valacyclovir Tablet
  Interventions: Drug: Valacyclovir
- Valtrex (Active Comparator): Reference Listed 1000 mg Valtrex Tablet
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — 1000 mg Tablet
  Arms: Valacyclovir
Drug: Valacyclovir — 1000 mg Tablet
  Other Names: Valtrex
  Arms: Valtrex

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of valacyclovir 1000 mg tablet (test) versus Valtrex (reference), administered as 1 x 1000 mg tablet under fasting conditions.

ELIGIBILITY:
Inclusion Criteria

* Male or female, non-smokers, 18 years of age and older.
* Capable of consent
* BMI greater than or equal to 19.0 and less than or equal to 30.0 kg/m2

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses or surgery within 4 weeks of the administration of study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol or drug abuse within one year prior to the screening visit
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40% alcohol]) or positive urine drug screen at screening.
* Use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, valacyclovir, acyclovir, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to the administration of the study medication.
* Use of an investigational drug or participation in an investigation study within 30 days prior to the administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 90 days preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, could contraindicate the subjects participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Intolerance to venipunctures.
* Clinically significant history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Unable to understand or unwilling to sign the Informed Consent Form.
* Breast-feeding.
* Positive serum pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception:
* Intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration),
* Condom or diaphragm + spermicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of drug substance in plasma) | Blood samples collected over 16 hour period
  Bioequivalence based on Cmax
AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) | Blood samples collected over 16 hour period
  Bioequivalence based on AUC0-t
AUC0-inf (area under the concentration-time curve from time zero to infinity) | Blood samples collected over 16 hour period
  Bioequivalence based on AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., East Grand Forks, Minnesota, United States